CLINICAL TRIAL: NCT00493883
Title: Use of TheraSphere® Yttrium-90 Glass Microspheres for Primary and Metastatic Liver Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Southwestern Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTCT 06-11
Record Dates: First submitted 2007-06-26; First posted 2007-06-28 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Carcinoma, Hepatocellular; Liver Neoplasms
Keywords: Therasphere; Yttrium; liver; cancer; radiation
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TheraSphere (Other): Y-90 is incorporated into very tiny glass beads, it can be injected into the liver through the blood vessels supplying the liver
  --------------------------------------------------------------------------------
  Interventions: Device: yttrium Y 90 microspheres (TheraSphere®)

INTERVENTIONS:
Device: yttrium Y 90 microspheres (TheraSphere®) — Y-90 is incorporated into very tiny glass beads, it can be injected into the liver through the blood vessels supplying the liver

SUMMARY:
The purpose of this study is to provide supervised access to treatment with TheraSphere® to eligible patients with primary and metastatic cancer and evaluate response to treatment, survival and toxicity.

The study has the following objectives:

* Provide supervised access to treatment with TheraSphere to eligible patients with primary and metastatic cancer to the liver.
* Evaluate patient experience and toxicities associated with TheraSphere treatment
* Evaluate predisposing factors that may influence results and toxicity

DETAILED DESCRIPTION:
This study will use angiographic administration of radioactive TheraSphere® Yttirum-90 microspheres into the hepatic artery, to treat 50 patients with primary or secondary cancer involving the liver. The study population are those who have failed standard therapies, have a majority of their cancer in the liver, have a good performance status and reasonable hepatic function. Outcomes being studied are response to treatment, survival and toxicity.

1. Range of patients who can be offered TheraSphere®
2. Tumor response rates, in terms of size, volume, contrast enhancement and PET avidity
3. Survival time
4. Determine response in relation to histology and other parameters
5. Ability to tolerate repeat treatments
6. Toxicity, which may include radiation induced liver damage, pain, consequences of shunting, toxic deaths.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18.
2. Cancer visible in liver on CT,MR,US or PET scan.
3. Primary cancer in the liver (hepatocellular carcinoma), or metastatic cancer involving the liver from a primary such as but not limited to lung, breast, colon, upper GI, neuroendocrine, melanoma.
4. Life expectancy greater than 2 months
5. Performance status of ECOG 2 or better (Ambulatory and capable of all selfcare, but unable to carry out any work activities. Up and about more than 50% of waking hours.)
6. Patients have tried and/or are aware of all FDA approved therapies for their condition.

Exclusion Criteria:

1. Vascular shunt that cannot be corrected.
2. Bulky cancer outside of liver. Active cancer within the liver should be a greater volume than the active cancer outside the liver / in the remainder of body.
3. Pregnancy
4. Hematologic primary such as lymphoma, leukemia, myeloma.
5. Body weight 300 lbs. and above
6. Evidence of portal hypertension, splenomegaly or ascites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2006-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Tumor response rates, in terms of size, volume, contrast enhancement and PET avidity | 2 to 3 months after treatment(s) up to 2 years
Toxicity, which may include radiation induced liver damage, pain, consequences of shunting, toxic deaths. | 2 years
Survival time | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: James P Flynn, MD, Principal Investigator — Southwestern Regional Medical Center
Locations (1):
- Cancer Treatment Centers of America at Southwestern Regional Medical Center, Tulsa, Oklahoma, United States

REFERENCES:
- [Background] Campbell AM, Bailey IH, Burton MA. Tumour dosimetry in human liver following hepatic yttrium-90 microsphere therapy. Phys Med Biol. 2001 Feb;46(2):487-98. doi: 10.1088/0031-9155/46/2/315. PMID 11229728
- [Background] Herba MJ, Thirlwell MP. Radioembolization for hepatic metastases. Semin Oncol. 2002 Apr;29(2):152-9. doi: 10.1053/sonc.2002.31672. PMID 11951213
- [Background] Wong CY, Salem R, Raman S, Gates VL, Dworkin HJ. Evaluating 90Y-glass microsphere treatment response of unresectable colorectal liver metastases by [18F]FDG PET: a comparison with CT or MRI. Eur J Nucl Med Mol Imaging. 2002 Jun;29(6):815-20. doi: 10.1007/s00259-002-0787-4. Epub 2002 Mar 29. PMID 12029557
- [Background] Goin JE, Salem R, Carr BI, Dancey JE, Soulen MC, Geschwind JF, Goin K, Van Buskirk M, Thurston K. Treatment of unresectable hepatocellular carcinoma with intrahepatic yttrium 90 microspheres: a risk-stratification analysis. J Vasc Interv Radiol. 2005 Feb;16(2 Pt 1):195-203. doi: 10.1097/01.RVI.0000142602.79459.90. PMID 15713920
- [Background] Murthy R, Xiong H, Nunez R, Cohen AC, Barron B, Szklaruk J, Madoff DC, Gupta S, Wallace MJ, Ahrar K, Hicks ME. Yttrium 90 resin microspheres for the treatment of unresectable colorectal hepatic metastases after failure of multiple chemotherapy regimens: preliminary results. J Vasc Interv Radiol. 2005 Jul;16(7):937-45. doi: 10.1097/01.RVI.0000161142.12822.66. PMID 16002501
- [Background] Wong CY, Qing F, Savin M, Campbell J, Gates VL, Sherpa KM, Lewandowski RJ, Nagle C, Salem R. Reduction of metastatic load to liver after intraarterial hepatic yttrium-90 radioembolization as evaluated by [18F]fluorodeoxyglucose positron emission tomographic imaging. J Vasc Interv Radiol. 2005 Aug;16(8):1101-6. doi: 10.1097/01.RVI.0000168104.32849.07. PMID 16105922
- [Background] Salem R, Lewandowski RJ, Atassi B, Gordon SC, Gates VL, Barakat O, Sergie Z, Wong CY, Thurston KG. Treatment of unresectable hepatocellular carcinoma with use of 90Y microspheres (TheraSphere): safety, tumor response, and survival. J Vasc Interv Radiol. 2005 Dec;16(12):1627-39. doi: 10.1097/01.RVI.0000184594.01661.81. PMID 16371529
- [Background] Lewandowski RJ, Thurston KG, Goin JE, Wong CY, Gates VL, Van Buskirk M, Geschwind JF, Salem R. 90Y microsphere (TheraSphere) treatment for unresectable colorectal cancer metastases of the liver: response to treatment at targeted doses of 135-150 Gy as measured by [18F]fluorodeoxyglucose positron emission tomography and computed tomographic imaging. J Vasc Interv Radiol. 2005 Dec;16(12):1641-51. doi: 10.1097/01.RVI.0000179815.44868.66. PMID 16371530
- [Background] Wong CY, Savin M, Sherpa KM, Qing F, Campbell J, Gates VL, Lewandowski RJ, Cheng V, Thie J, Fink-Bennett D, Nagle C, Salem R. Regional yttrium-90 microsphere treatment of surgically unresectable and chemotherapy-refractory metastatic liver carcinoma. Cancer Biother Radiopharm. 2006 Aug;21(4):305-13. doi: 10.1089/cbr.2006.21.305. PMID 16999596
- [Background] Salem R, Thurston KG. Radioembolization with yttrium-90 microspheres: a state-of-the-art brachytherapy treatment for primary and secondary liver malignancies: part 3: comprehensive literature review and future direction. J Vasc Interv Radiol. 2006 Oct;17(10):1571-93. doi: 10.1097/01.RVI.0000236744.34720.73. PMID 17056999
- [Background] Sato K, Lewandowski RJ, Bui JT, Omary R, Hunter RD, Kulik L, Mulcahy M, Liu D, Chrisman H, Resnick S, Nemcek AA Jr, Vogelzang R, Salem R. Treatment of unresectable primary and metastatic liver cancer with yttrium-90 microspheres (TheraSphere): assessment of hepatic arterial embolization. Cardiovasc Intervent Radiol. 2006 Jul-Aug;29(4):522-9. doi: 10.1007/s00270-005-0171-4. PMID 16729228